CLINICAL TRIAL: NCT00004382
Title: Phase II Study of Tin Mesoporphyrin vs Phototherapy for Hyperbilirubinemia in Premature Newborns
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: Rockefeller University (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 199/12022; RUH-0330795B
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2008-09-09 (Estimated); Status verified 2008-09

CONDITIONS: Hyperbilirubinemia
Keywords: hematologic disorders; hyperbilirubinemia; rare disease
MeSH Terms: conditions — Hyperbilirubinemia; Hematologic Diseases; Rare Diseases | interventions — tin mesoporphyrin; Phototherapy

INTERVENTIONS:
Drug: tin mesoporphyrin
Procedure: Phototherapy

SUMMARY:
OBJECTIVES: I. Compare the effectiveness of a single dose of tin mesoporphyrin and special blue light phototherapy in controlling hyperbilirubinemia in premature newborns in Greece.

II. Evaluate the dose of tin mesoporphyrin sufficient to alleviate the need for phototherapy without adverse effects in these newborns.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients are randomly assigned to a clinical group within 96 hours of birth. Patients are stratified by gestational age, clinical status, and age at treatment.

One group receives tin mesoporphyrin. Patients are crossed to phototherapy if the plasma bilirubin concentration reaches the treatment threshold.

The second group receives phototherapy with Special Blue fluorescent lamps for at least 24 hours. Patients receive a second phototherapy course if the plasma bilirubin concentration reaches the treatment threshold within 24 hours of the first course.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Premature infants of gestational age 210 to 251 days
* No blood group isoimmunization (direct Coombs' positive), e.g., rhesus or ABO
* No glucose-6-phosphate dehydrogenase deficiency

--Prior/Concurrent Therapy--

* No maternal phenobarbital in last month of pregnancy

--Patient Characteristics--

Renal: No congenital renal abnormality

Cardiovascular: No congenital heart abnormality

Pulmonary: No asphyxia requiring assisted ventilation at delivery

Other: No other major congenital abnormality, i.e.:

* Central nervous system
* Chromosomal
* Gastrointestinal

No evident or suspected congenital infection, i.e.:

* Cytomegalovirus
* Herpes
* Rubella
* Syphilis

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80
Dates: Start 1999-12; Primary Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Attallah Kappas, Study Chair — Rockefeller University